CLINICAL TRIAL: NCT00736411
Title: IVF and Acupuncture for Infertility: A Randomized Controlled Trail
Brief Title: In Vitro Fertilization (IVF) and Acupuncture for Infertility
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Adjustments to ensure clear outcomes and scientific merit integrated. Study closed at 14 subjects. New protocol submitted to IRB.
Sponsor: Pacific Fertility Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28.005-2
Record Dates: First submitted 2008-08-13; First posted 2008-08-15 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Infertility
Keywords: infertility; IVF; acupuncture
MeSH Terms: conditions — Infertility | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): IVF
  Interventions: Procedure: IVF
- II (Other): treatment
  Interventions: Procedure: acupuncture

INTERVENTIONS:
Procedure: acupuncture — 16 treatments over 8 weeks
  Arms: II
Procedure: IVF — one 4 week IVF cycle
  Arms: 1

SUMMARY:
The aim of this investigation is to determine the value of combining acupuncture with infertility patients undergoing In Vitro Fertilization (IVF). The investigators will measure the outcomes of endometrial lining, uterine blood flow, hormones, stress levels, and pregnancy and live birth rates.

ELIGIBILITY:
Inclusion Criteria:

* females between 21 and 42 years old
* primary or secondary infertility
* no more than 2 previously failed IVF cycles
* undergoing IVF
* FSH < 11

Exclusion Criteria:

* FSH > 11
* using an egg donor
* using PGD
* using heparin or lovanox protocols
* estradiol level less than 20 or over 80
* taking herbal therapy

Ages: 21 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
pregnancy | week 10 of study

SECONDARY OUTCOMES:
uterine blood flow | final measurement in week 8

CONTACTS AND LOCATIONS:
Overall Officials: Caylie J See, L.Ac., Study Director — Pacific Fertility Center
Locations (1):
- Pacific Fertility Center, San Francisco, California, United States